CLINICAL TRIAL: NCT05671185
Title: Therapeutic Effect of Repetitive Transcranial Magnetic Stimulation for Depressive, Positive and Negative Symptoms, and Physiological Indices of Schizophrenia Patients
Brief Title: rTMS for Depressive, Positive and Negative Symptoms, and Physiological Indices of Schizophrenia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202210011DINC
Record Dates: First submitted 2022-12-18; First posted 2023-01-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- conventional rTMS (Experimental): target: left DLPFC
  protocol: 10Hz for 4 seconds, 120% motor threshold, 75 trains with 26-second interval, 3000 pulses per session, one session per day, five sessions per week, two weeks in total
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- iTBS (Experimental): target: left DLPFC
  protocol: 3 pulses at 50Hz, 90% motor threshold, repeated at 5Hz, 60 trains of 10 bursts with 8-second intervals, 1800 pulses per session, one session per day, five sessions per week, two weeks in total
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- sham rTMS (Sham Comparator): target: left DLPFC
  sham probe, the same protocol as active conventional rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- sham iTBS (Sham Comparator): target: left DLPFC
  sham probe, the same protocol as active iTBS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS using Magstim TMS system is delivered at the left dorsolateral prefrontal cortex

SUMMARY:
Around 40% of schizophrenia patients present depressive symptoms, which are associated with elevated suicide and violence risk and poor prognosis and quality of life. Recent meta-analysis showed the effect size of antidepressants for depressive symptoms of schizophrenia patients was as low as 0.25, so new therapeutic approach is warranted.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, anesthesia-free brain stimulation therapy for treatment refractory depression. Currently, rTMS is classified as high-frequency stimulation (>5Hz, usually 10Hz or 20Hz) and low-frequency inhibition (usually 1Hz). Intermittent theta burst stimulation (iTBS) is a new variant of rTMS, with stimulation frequency as high as 50Hz. Compared with high-frequency rTMS, iTBS has similar therapeutic effect and shorter stimulation duration. Up to now, studies exploring treatment effect of rTMS or iTBS for schizophrenia patients mainly focused on negative symptoms rather than depressive symptoms. Therefore, this study aims to explore treatment effect of rTMS or iTBS of depressive symptoms, negative symptoms, cognitive function and physiological indices for schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Able to give informed consent
* Diagnosed with schizophrenia or schizoaffective disorder according to DSM-5
* Has a score ≥ 7 on Calgary depression scale for schizophrenia
* The principal psychotropic agents are not changed within one month of the first session of rTMS

Exclusion Criteria:

* DSM-5 defined substance use disorder (excluding tobacco) in the past 3 months
* Have clinically relevant cognitive impairment (e.g., delirium, intellectual disability or MMSE < 15)
* With electronic and/or magnetic implants (e.g. pacemaker, implantable cardioverter defibrillator [ICD], cerebral shunts, cochlear implant, etc.)
* With metallic or mechanic fragments (e.g., screws, plates, stents, clips, etc.)
* Pregnant, or has a pregnancy plan within 3 months
* With any known or history of neurological conditions including cerebral vascular accidents, epilepsy (or epileptiform waves detected by EEG prior to the first session of rTMS), brain tumor or space occupying lesion
* Received rTMS or iTBS treatment within 3 months
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Calgary Depression Scale for Schizophrenia | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  A 9-item scale developed for detecting major depressive episode for schizophrenia patients. Total score ranges from 0 to 27. Lower score indicates less depressive symptoms. A cut-off of 7 points yields to sensitivity of 85% and specificity of 82%.

SECONDARY OUTCOMES:
Change from Baseline in Positive and Negative syndrome scale | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  A 30-item scale developed to evaluating positive, negative and general symptoms for schizophrenia patients. Total score ranges from 30 to 210. Lower score indicates fewer schizophrenic symptoms.
Change from Baseline in Negative symptoms assessment 16 | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  A scale developed to evaluating negative symptoms for schizophrenia patients. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 domain scores are the sum of item scores in each domain i.e. communication (min score 4, max score 24), emotion/affect (min 3, max 18), social involvement (min 3, max 18), motivation (min 4, max 24), and retardation (min 2, max 12); with higher scores denoting more severe negative symptoms in schizophrenia.
Change from Baseline in Clinical global impression | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  A scale for primary-care psychiatrist to evaluate global symptom severity of a patient in comparison with others with same diagnosis. Lower score indicates less severe illness.
Change from Baseline in Self-Reported Graphic version of the Personal and Social Performance Scale | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  A 22-item self-rated scale for schizophrenia patients, which includes four domains, i.e., global function (6 items, total scores 6-18), personal and social performance (5 items, total scores 5-15), self-care (6 items, total scores 6-18) and disturbing behaviors (5 items, total scores 5-15). Lower score indicates less severe illness.

OTHER OUTCOMES:
Change from Baseline in Physiological Parameters - Heart Rate Variability | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  Measurement of parasympathetic activity.
Change from Baseline in Physiological Parameters - Skin Conductance | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  Measurement of sympathetic activity.
Change from Baseline in Physiological Parameters - Body Temperature | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  Measurement of autonomic nervous system.
Change from Baseline in Physiological Parameters - Respiratory Rate | baseline (Day 1), Day 8, Day 15, Day 29, Day 57, Day 85
  Measurement of autonomic nervous system.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hao Ma, MD, Principal Investigator — Department of Psychiatry, National Taiwan University Hospital Yunlin Branch
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin, Taiwan